CLINICAL TRIAL: NCT05290090
Title: Prospective, Single-arm, Phase II Clinical Study of Rituximab, Lenalidomide, and Zanubrutinib Combination Regimen Followed by Immunochemotherapy in the Treatment of Elderly Patients With Newly-diagnosed Diffuse Large B-cell Lymphoma
Brief Title: ZR2 Followed by Immunochemotherapy in Elderly Patients With Newly-diagnosed DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZR2+RCHOP
Record Dates: First submitted 2022-01-28; First posted 2022-03-22 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: diffuse large B cell lymphoma; elderly; rituximab; lenalidomide; zanubrutinib; treatment; chemo-free
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Lenalidomide; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab, lenalidomide, zanubrutinib and RCHOP (Experimental): Rituximab, lenalidomide, zanubrutinib for 2 cycles: rituximab 375mg/m2, d1, lenalidomide 10mg qd d1-10, zanubrutinib 160mg bid.
  RCHOP for 4 cycles: rituximab 375mg/m2 d0, cyclophosphamide: 750mg/m2 d1, epirubicin: 75mg/m2 d1 (or liposomal doxorubicin 35mg/m2 d1), vindesine 4mg d1, prednisone: 100mg, d1-5.
  Interventions: Drug: Rituximab, Lenalidomide, Zanubrutinib and RCHOP

INTERVENTIONS:
Drug: Rituximab, Lenalidomide, Zanubrutinib and RCHOP — chemo free period (21 days as a cycle, a total of 2 cycles): rituximab 375mg/m2, d1, lenalidomide 10mg qd d1-10, zanubrutinib 160mg bid.
  Immunochemotherapy period: RCHOP regimen (21 days as 1 cycle, a total of 4 cycles): rituximab 375mg/m2 d0, cyclophosphamide: 750mg/m2 d1, epirubicin: 75mg/m2 d1 (or liposomal doxorubicin 35mg/m2 d1), vindesine 4mg d1, prednisone: 100mg, d1-5.
  Other Names: BGB-3111

SUMMARY:
As the most common subtype of lymphoma, diffuse large B-cell lymphoma (DLBCL) is an aggressive but potentially curable malignancy. The poor prognosis of elderly DLBCL patients may be related to the biological behavior of the disease, more comorbidities, poor performance status, and inability to tolerate standard-intensity immunochemotherapy. The investigators plan to use ZR2 regimen(rituximab, lenalidomide and zanubrutinib) for 2 cycles followed by immunochemotherapy for up to 4 cycles in elderly newly diagnosed DLBCL patients.

DETAILED DESCRIPTION:
DLBCL mostly occurs in the elderly, with a median age at diagnosis of 66 years. Age over 60 years is a poor prognostic factor for DLBCL and is included in the International Prognostic Index (IPI) to stratify patients for prognosis. So there is an unmet need for treatment in this population. Both lenalidomide and BTK inhibitor single drugs have shown certain efficacy in DLBCL patients, and many studies have also explored the effectiveness of rituximab, lenalidomide and BTK inhibitor combination regimen in the treatment of DLBCL. Therefore, the investigators plan to use ZR2 regimen(rituximab, lenalidomide and zanubrutinib) for 2 cycles to reduce tumor burden, improve the patient's physical condition, and improve the tolerance to immunochemotherapy in elderly newly diagnosed DLBCL patients. Up to 4 cycles of immunochemotherapy were then administered sequentially in order to reduce the overall chemotherapy intensity of the patients and improve the long-term quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participate in the clinical study voluntarily: fully understand and be informed of the study and sign the informed consent in person; Willing to follow and be able to complete all test procedures.
2. Age: 70-85 years old, or 65-70 years old with ECOG score ≥2 points, both male and female.
3. Histopathologically confirmed as diffuse large B-cell lymphoma, not otherwise specified.
4. No prior anti-tumor therapy, such as chemotherapy, radiotherapy, immunotherapy or biotherapy (tumor vaccine, cytokine, or anti-tumor growth factor).
5. At least one evaluable or measurable lesion that meets Lugano2014 criteria (evaluable lesion: PET/CT examination showing increased uptake in lymph nodes or extranodal areas (higher than liver) and PET/CT and/or CT consistent with lymphoma; Measurable lesions: nodular lesions >15mm in length or extragendal lesions >10mm in length with increased FDG uptake).
6. Adequate organ and bone marrow function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function and immune deficiency (no blood transfusion, granulocytic colony stimulating factor or other relevant medical support within 14 days prior to the use of the study drug) :

   1. neutrophil absolute count (ANC) ≥1.5×109/L (1500/mm3), platelet ≥75×109/L, hemoglobin ≥100g/L (if bone marrow is involved, platelet ≥50×109/L, ANC ≥1.0×109/L, hemoglobin ≥80g/L).
   2. Liver function: serum bilirubin ≤2.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal value (AST or ALT≤5 times the upper limit of normal value is allowed if liver is involved).
   3. Renal function: creatinine clearance ≥60 mL/min (estimated according to the Cockcroft-Gault formula).
   4. Coagulation function: INR≤1.5 times the upper limit of normal value; PT and APTT≤1.5 times the upper limit of normal value.
7. Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.
8. Negative serum pregnancy test and effective contraceptive use from signing informed consent until 6 months after the last chemotherapy.
9. Life expectancy > 3 months.

Exclusion Criteria:

1. Pathological subtypes: primary central nervous system diffuse large B-cell lymphoma, primary mediastinal large B-cell lymphoma, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement, high-grade B-cell lymphoma, not otherwise specified. EBV positive diffuse large B-cell lymphoma
2. Hemophagocytic syndrome at the time of diagnosis.
3. Central nervous system involvement secondary to lymphoma.
4. Participating in other clinical studies.
5. Medical history of other active malignancy within 2 years prior to enrollment, except for the following conditions:(1) adequately treated in situ of the cervix carcinoma; (2) local basal cell carcinoma or squamous cell carcinoma of skin; (3) Pre-existing malignant disease that is under control and has undergone local radical treatment (surgical or other forms).
6. History of Human Immunodeficiency Virus (HIV) infection and/or acquired Immunodeficiency syndrome. Patients with positive hepatitis B surface antigen or hepatitis C virus antibody must be tested hepatitis B virus DNA (no more than 1000 iu/ml) and HCV RNA detection (below the detection limit). Patients with hepatitis B virus carriers, or stabilized hepatitis B with anti-virus treatment and cured hepatitis C can be included.
7. Major surgery was performed within 28 days prior to study initiation.
8. Any active infection, including bacterial, fungal or viral infections, that requires systemic antiinfection therapy within 14 days prior to treatment.
9. Accompanied with severe or uncontrolled disease, including symptomatic of congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer or A history of severe hemorrhagic diseases, such as hemophilia A, hemophilia B, von willebrand disease or blood transfusion or other medical intervention history of spontaneous bleeding.
10. History of stroke or intracranial hemorrhage within 6 months prior to first administration of the study drug.
11. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months.
12. Patients who must take antiplatelet drugs and anticoagulants at the same time due to underlying diseases, and there is no alternative treatment plan.
13. Continuous treatment with strong and moderate CYP3A inhibitors or CYP3A inducers is required. Patients were excluded if they had taken a CYP3A potent or moderate-acting inhibitor or inducer within 7 days prior to the first administration of the study drug (or had taken these drugs for less than 5 half-lives).
14. Hypersensitivity to the experimental drug is known.
15. Patients deemed unsuitable for the study by researchers.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 21days after the end of treatment
  overall response rate

SECONDARY OUTCOMES:
PFS | From date of first day of treatment until the date of first documented progression, assessed up to 24 months
  Progression Free Survival
OS | From date of first day of treatment until the date of first documented date of death from any cause, assessed up to 24 months
  Overall Survival
AE and SAE | From date of first day of treatment until 30 day after last treatment
  Adverse event and serious adverse event
Performance status | At screening period, after 2 cycles of ZR2 regimen(each cycle is 21 days), after 2 cycles of RCHOP regimen(each cycle is 21 days) and 21days after the end of treatment
  Assess the patient's performance status according to the Barthel index. Patients will be classified into 5 scales with the score ranging from 0 to 100: 0-20 points=extremely severe functional impairment; 25-45 points=severe functional impairment; 50-70 points=moderate functional impairment; 75-95 points=mild functional impairment; 100 points=normal. Higher scores mean a better outcome.
Life quality | At screening period, after 2 cycles of ZR2 regimen(each cycle is 21 days), after 2 cycles of RCHOP regimen(each cycle is 21 days) and 21days after the end of treatment
  Assess the patient's quality of life according to the EORTC QLQ-C30 questionnaire. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Yang, Principal Investigator — Zhejiang Cancer Hospital, Hangzhou, China
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No